CLINICAL TRIAL: NCT04463771
Title: An Umbrella Study of INCMGA00012 Alone and in Combination With Other Therapies in Participants With Advanced or Metastatic Endometrial Cancer Who Have Progressed on or After Platinum-Based Chemotherapy (POD1UM-204)
Brief Title: Safety and Efficacy of Retifanlimab (INCMGA00012) Alone or in Combination With Other Therapies in Participants With Advanced or Metastatic Endometrial Cancer Who Have Progressed on or After Platinum-based Chemotherapy.
Acronym: POD1UM-204
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Collaborators: GOG Foundation (Network); European Network of Gynaecological Oncological Trial Groups (ENGOT) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCMGA 0012-204; 2022-502600-79-00 (Registry Identifier: EU CT Number); 2020-000496-20 (EudraCT Number)
Expanded Access: NCT06910137 (Available)
Record Dates: First submitted 2020-07-06; First posted 2020-07-09 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Endometrial Cancer
Keywords: Endometrial Carcinoma; Endometrium Cancer; Neoplasms Endometrial; Advanced; Metastatic; PD-1; PD-L1; retifanlimab; INCMGA0012; INCAGN02385; INCAGN02390; PODIUM; LAG-3; TIM-3
MeSH Terms: conditions — Endometrial Neoplasms; Neoplasm Metastasis | interventions — epacadostat; pemigatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Group A - retifanlimab (Experimental): Select participants naïve to checkpoint inhibitors will be administered retifanlimab intravenously
  Interventions: Drug: retifanlimab
- Group B - retifanlimab (Experimental): Select participants naïve to checkpoint inhibitors will be administered retifanlimab intravenously
  Interventions: Drug: retifanlimab
- Group C - retifanlimab + epacadostat (Experimental): Select participants who are allowed on prior checkpoint inhibitors will be administered retifanlimab intravenously in combination with oral epacadostat (IDO1 inhibitor)
  Interventions: Drug: retifanlimab; Drug: epacadostat
- Group D - retifanlimab + pemigatinib (Experimental): Select participants who are allowed on prior checkpoint inhibitors will be administered retifanlimab intravenously in combination with oral pemigatininb (FGFR 1,2,3 inhibitor)
  Interventions: Drug: retifanlimab; Drug: pemigatinib
- Group E - retifanlimab + epacadostat (Experimental): Select participants naïve to checkpoint inhibitors will be administered retifanlimab intravenously in combination with oral epacadostat
  Interventions: Drug: retifanlimab; Drug: epacadostat
- Group F - retifanlimab + INCAGN02385 and INCAGN02390 (Experimental): Select participants who are allowed on prior checkpoint inhibitors will be administered retifanlimab in combination with INCAGN02385 and INCAGN02390 intravenously
  Interventions: Drug: INCAGN02385; Drug: INCAGN02390

INTERVENTIONS:
Drug: retifanlimab — INCMGA00012 administered intravenously on Day 1 of each 28-day cycle for up to 26 cycles.
  Other Names: INCMGA00012
  Arms: Group A - retifanlimab; Group B - retifanlimab; Group C - retifanlimab + epacadostat; Group D - retifanlimab + pemigatinib; Group E - retifanlimab + epacadostat
Drug: epacadostat — epacadostat will be administered orally BID.
  Arms: Group C - retifanlimab + epacadostat; Group E - retifanlimab + epacadostat
Drug: pemigatinib — pemigatinib will be administered orally QD.
  Arms: Group D - retifanlimab + pemigatinib
Drug: INCAGN02385 — INCAGN2385 will be administered every 2 weeks
  Arms: Group F - retifanlimab + INCAGN02385 and INCAGN02390
Drug: INCAGN02390 — INCAGN2390 will be administered every 2 weeks
  Arms: Group F - retifanlimab + INCAGN02385 and INCAGN02390

SUMMARY:
This is a multicenter, open-label, nonrandomized, Phase 2 umbrella study of retifanlimab in participants who have advanced or metastatic endometrial cancer that has progressed on or after platinum-based chemotherapy. retifanlimab will be administered as monotherapy or in combination with other immunotherapy or targeted agents.

ELIGIBILITY:
Inclusion Criteria:

* Ability to comprehend and willingness to sign a written ICF for the study. Note for Germany: This excludes individuals who are housed in an institution due to official or court order Women 18 years of age or older (or as applicable per local country requirements).
* Histologically confirmed diagnosis of advanced or metastatic endometrial cancer with disease progression on or after treatment with at least 1 platinum-containing regimen for advanced or metastatic disease.
* Groups A, B, and E: Have not been previously treated with a PD-(L)1 inhibitor.
* Group A only: Tumor tissue tested as MSI-High
* Group B only: Tumor tissue tested as deficient MMR or an ultra-mutated POLE tumor.
* Group D only: Tumor tissue tested as having an FGFR 1,2,3 mutation or alteration characterized as per protocol.
* Group E: Tumor tissue tested as MSS and PD-L1 positive.
* Group F: Radiological evidence of disease progression on or after prior PD (L)1 therapy and Tumor tissue tested as MSI-H
* Must have at least 1 measurable tumor lesion per RECIST v1.1.
* Willing to provide tumor tissue sample (fresh or archived).
* ECOG performance status 0 to 1.
* Willingness to avoid pregnancy.

Exclusion Criteria:

* Group A, B and E only: Histologically confirmed diagnosis of carcinosarcoma of the uterus.
* Histologically confirmed diagnosis of sarcoma of the uterus.
* Has disease eligible for potentially curative treatment.
* Receipt of anticancer therapy within 28 days of the first administration of study treatment, with the exception of localized radiotherapy.
* Toxicity of prior therapy that has not recovered to ≤ Grade 1 or baseline unless approved by the medical monitor.
* Groups C, D and F (combinations): limiting immune-related toxicity during prior checkpoint inhibitor therapy.
* Group F only: Previous treatment with LAG-# or TIM-3 therapy or lenvatinib; multiple metastases that achieved mixed tumor response to prior anti-PD-(L)1 therapy
* Has an active autoimmune disease requiring systemic immunosuppression with corticosteroids (> 10 mg/day of prednisone or equivalent) or immunosuppressive drugs within 14 days before the first dose of study treatment.
* Receiving chronic systemic steroids (> 10 mg/day of prednisone or equivalent):
* Known active CNS metastases and/or carcinomatous meningitis.
* Has known active hepatitis B or C.
* Has received a live vaccine within 28 days of the planned start of study treatment.
* Evidence of interstitial lung disease or active, noninfectious pneumonitis.
* Participants who are known to be HIV-positive with some protocol exceptions.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 206 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2026-04-14 (Estimated); Study Completion 2026-07-10 (Estimated)

PRIMARY OUTCOMES:
Group A - Objective Response Rate | up to 2.5 years
  Defined as the proportion of participants having a CR or PR according to RECIST v1.1, as assessed by Independent Central Review committee

SECONDARY OUTCOMES:
Group A -Duration of Response | up to 2.5 years
  Defined as the time from the first documented objective response (CR or PR) according to RECIST v1.1 (as determined by ICR) until disease progression or death due to any cause.
Group A - Disease Control Rate | up to 2.5 years
  Defined as the proportion of participants with CR, PR, or SD (as determined by ICR) as best response.
Group A - Overall Survival | up to 3.5 years
  Defined as the time from the first dose of study treatment until death due to any cause.
Group A - Progression Free Survival | up to 3.5 years
  Defined as the time from the first dose of study treatment until disease progression (as determined by ICR) or death due to any cause.
Group B -Duration of Response | up to 2.5 years
  Defined as the time from the first documented objective response (CR or PR) according to RECIST v1.1 (as determined by ICR) until disease progression or death due to any cause.
Group B - Disease Control Rate | up to 2.5 years
  Defined as the proportion of participants with CR, PR, or SD (as determined by ICR) as best response.
Group B - Overall Survival | up to 3.5 years
  Defined as the time from the first dose of study treatment until death due to any cause.
Groups B - Objective Response Rate | up to 2 years
  Defined as the proportion of participants having a CR or PR according to RECIST v1.1, as assessed by Independent Central Review committee
Group B - Progression Free Survival | up to 3.5 years
  Defined as the time from the first dose of study treatment until disease progression (as determined by ICR) or death due to any cause.
Groups C, D, E and F - Objective Response Rate | up to 2 years
  Defined as the proportion of participants having a CR or PR according to RECIST v1.1, as assessed by Independent Central Review committee
Number of Treatment-Related Adverse Events | up to 4 years
  Adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug/treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Cornfield, Study Director — Incyte Corporation
Locations (65):
- United States (29):
  - Alaska Womens Cancer Care Akwcc, Anchorage, Alaska
  - Honorhealth, Phoenix, Arizona
  - Arizona Oncology Associates, Tucson, Arizona
  - UCLA Medical Hematology & Oncology, Los Angeles, California
  - Olive View Med Ctr, Sylmar, California
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Miami Cancer Institute, Miami, Florida
  - Mount Sinai Medical Center Comprehensive Cancer Center, Miami Beach, Florida
  - Advent Health Medical Group-Orlando 2501, Orlando, Florida
  - H. Lee Moffitt Cancer Center and Research Institute Hospital, Tampa, Florida
  - Georgia Cancer Center, Augusta, Georgia
  - Barbara Ann Karmanos Cancer Hospital, Detroit, Michigan
  - Minnesota Oncology-Maplewood, Coon Rapids, Minnesota
  - Midwest Cancer Care, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - New Mexico Cancer Care Alliance, Albuquerque, New Mexico
  - Laura & Isaac Perlmutter Cancer Ctr, New York, New York
  - University of North Carolina At Chapel Hill, Chapel Hill, North Carolina
  - The Ohio State University Wexner Medical Center Division of Gynecologic Oncology, Hilliard, Ohio
  - Willamette Valley Cancer Institute, Eugene, Oregon
  - Texas Oncology-Tyler, Sioux Falls, South Dakota
  - Tennessee Oncology, Nashville, Tennessee
  - Texas Oncology-Austin Center, Austin, Texas
  - Texas Oncology-Fort Worth South Henderson, Fort Worth, Texas
  - Texas Oncology San Antonio, San Antonio, Texas
  - Texas Oncology the Woodlands, Shenandoah, Texas
  - Virginia Commonwealth University, Richmond, Virginia
- Belgium (6):
  - O.L.V Ziekenhuis, Aalst
  - Institut Jules Bordet, Brussels
  - Ghent University Hospital, Ghent
  - Universitaire Ziekenhuis Leuven - Gasthuisberg, Leuven
  - Centre Hospitalier Universitaire de Liege - Sart Tilman, Liège
  - Chu Ucl Namur de Saint Elisabeth, Namur
- France (6):
  - Chu Besancon Hospital Jean Minjoz, Besançon
  - Institut Bergonie, Bordeaux
  - Hospital Cochin Cancerologie, Paris
  - Cario - Centre Armoricain de Radiotherapie Imagerie Medicale Et Oncologie, Plérin
  - Centre de Lutte Contre Le Cancer - Institut de Cancerologie de L'Ouest - Rene Gauducheau, Saint-Herblain
  - Institut Gustave Roussy, Villejuif
- Georgia (6):
  - High Technology Hospital Medcenter, Batumi
  - Jsc Evex Hospitals, Kutaisi
  - Todua Clinic, Llc, Tbilisi
  - Caucasus Medical Centre Llc, Tbilisi
  - INNOVA, Tbilisi
  - Multiprofile Clinic Consilium Medulla Llc, Tbilisi
- Germany (4):
  - Charite - Campus Virchow-Klinikum, Berlin
  - University Clinic Carl Gustav Carus Technical University Dresden, Dresden
  - Klinikum Kassel Gmbh, Kassel
  - Universitarsfrauenklinik Ulm, Ulm
- Greece (4):
  - Alexandra General Hospital of Athens, Athens
  - University Hospital of West Attica - Attikon, Athens
  - Hygeia Hospital, Marousi
  - Euromedica General Clinic of Thessaloniki, Thessaloniki
- Italy (10):
  - Azienda Ospedaliero-Universitaria Di Bologna Policlinico S. Orsola - Malpighi, Bologna
  - Presidio Ospedaliero Di Summa Antonio Perrino, Brindisi
  - Istituto Scientifico Romagnolo Per Lo Studio E La Cura Dei Tumori, Meldola
  - Istituto Di Ricovero E Cura A Carattere Scientifico (Irccs) Ospedale San Raffaele, Milan
  - Comitato Etico Fondazione Irccs Istituto Nazionale Dei Tumori Milano, Milan
  - European Institute of Oncology, Milan
  - Istituto Nazionale Tumori Irccs Fondazione Pascale, Napoli
  - Iov - Istituto Oncologico Veneto Irccs, Padua
  - Fondazione Policlinico Universitario Agostino Gemelli Irccs, Roma
  - Ospedale Santa Maria Ca Foncello, Treviso

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- See also: Safety and Efficacy of Retifanlimab (INCMGA00012) Alone or in Combination With Other Therapies in Participants With Advanced or Metastatic Endometrial Cancer Who Have Progressed on or After Platinum-based Chemotherapy. — https://incyteclinicaltrials.com/studies/incmga-0012-204